CLINICAL TRIAL: NCT07076563
Title: Chronic Effects of Ice Cream Enriched With Cimarrón Bean Extrudate on Metabolic and Cardiovascular Risk Markers: A Randomized Crossover Clinical Trial in Adults
Brief Title: Ice Cream Enriched With Cimarrón Bean Extrudate and Cardiovascular Risk in Adults
Acronym: ICE-CBE-CARD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Collaborators: Centro de Estudios en Alimentos Procesados (Other)
Responsible Party: Principal Investigator, Iván Palomo González, Principal Investigator, University of Talca
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CH-HEP-UTALCA-F29-2021
Record Dates: First submitted 2025-06-25; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Risk Factors; Insulin Resistance; Overweight (BMI > 25)
Keywords: Phaseolus vulgaris; Funtional food; Legume-base food; cardiovascular disease; cardiovascular risk
MeSH Terms: conditions — Insulin Resistance; Overweight; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind, crossover clinical trial with two arms: one receiving a functional ice cream enriched with 10 g of Cimarrón bean extrudate (intervention) and one receiving a placebo ice cream (control), both matched for appearance and taste. Participants are randomly assigned to one of two groups (Alfa or Gamma).
  Each participant undergoes two intervention phases, each lasting four weeks, separated by washout period. The order of receiving the intervention or placebo is randomized. During each intervention period, participants consume 100 g/day of the assigned ice cream. Fasting blood samples and anthropometric data are collected at the beginning and end of each phase.
  Randomization is performed using block randomization stratified by sex, age, and body mass index (BMI), to ensure balance across treatment sequences.
  This crossover model allows each participant to serve as their own control, reducing inter-individual variability and increasing statistical power
Who Masked: Participant
Masking Description: Participants were blinded to the intervention type (placebo vs. functional ice cream) by providing both ice creams with identical appearance, texture, and flavor.
  The investigators were not blinded due to the need to manage logistics and sample handling. However, participants were unaware of their group assignment to minimize bias in self-reported adherence and perception of effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Ice Cream (Placebo Comparator): Participants consume 100 g/day of placebo ice cream for 4 weeks. The placebo ice cream is organoleptically identical to the intervention but does not contain Cimarrón bean extrudate. After a washout period, participants cross over to the intervention arm.
  Interventions: Dietary Supplement: Placebo Ice Cream
- Functional Ice Cream Enriched with Cimarrón Bean Extrudate (Experimental): Participants consume 100 g/day of ice cream enriched with 10 g of Cimarrón bean extrudate for 4 weeks. After a washout period, participants cross over to the placebo arm.
  Interventions: Dietary Supplement: Functional Ice Cream with Cimarrón Bean Extrudate

INTERVENTIONS:
Dietary Supplement: Functional Ice Cream with Cimarrón Bean Extrudate — Ice cream containing 10 g of Cimarrón bean extruded (Phaseolus vulgaris L., local variety "Cimarrón") 100 g per portion. Participants consume 100 g daily (two 50 g portions, ~2 hours after a main meal) for 4 weeks.
  Arms: Functional Ice Cream Enriched with Cimarrón Bean Extrudate
Dietary Supplement: Placebo Ice Cream — Ice cream without Cimarrón bean extrudate, matched in appearance, taste, and texture to the functional ice cream. Participants consume 100 g daily (two 50 g portions) for 4 weeks.
  Arms: Placebo Ice Cream

SUMMARY:
The goal of this clinical trial is to evaluate the chronic effects of consuming a functional ice cream enriched with Cimarrón bean (Phaseolus vulgaris local variety Cimarrón) extrudate in adults with at least one cardiovascular risk factor.

The main question it aims to answer is:

* Does chronic daily consumption of the functional ice cream with Cimarrón bean extrudate improve fasting glucose, insulin, lipid profile, and other cardiovascular risk markers?

Researchers will compare a functional ice cream containing 10 g of extrudate per100 g to a placebo version without extrudate, using a crossover design in which participants consume both versions for 4 weeks each, separated by a 3-week washout period to determine metabolic responses.

Participants will:

* Attend clinical visits in fasting conditions at the beginning and end of each 4-week intervention to provide blood samples for glucose, insuli, lipid profile, complete blood count plus Erythrocyte sedimentation rate and HbA1c assessment.
* Undergo anthroprometric measurements and blood pressure assessment at the beginning and end of each 4-week intervention.
* Consume 100g/day of the assigned ice cream during each phase (Two phases)

DETAILED DESCRIPTION:
This randomized, single-blind, crossover clinical trial assesses the effects of daily consumption of a functional ice cream enriched with Cimarrón bean extrudate (Phaseolus vulgaris L., local variety Cimarrón) extrudate in adults with at least one cardiovascular risk factor.

Eligible participants are adults (20-59 years) health or present at least one cardiovascular risk factor (e.g., smoking, insulin resistance, overweight/obesity, hypertension) and a BMI between 18.5 and 39.9 kg/m^2.

Participants are randomized into two groups (Alfa and Gamma) to receive either the placebo or functional ice cream first. Each intervention period lasts 4 week during which participants consume 100 g/day of the assigned ice cream (two 50 g portions, ~2 hours after a main meal). Following a 3-week washout period, participants switch to the alternate intervention. At the beginning and end of each intervention period, anthropometric assessments are performed, including body weight, height, body mass index (BMI), waist circumference, and mid-upper arm circumference. Additionally, fasting blood samples are collected to assess glucose, insulin, lipid profile, complete blood count plus erythrocyte sedimentation rate, HbA1c, and blood pressure.

The placebo or functional ice cream are organoleptically identical to ensure blinding. Randomization is stratified by sex, age, and BMI using balanced block randomization with R software (v4.5.0).

The primary outcomes are the within-subject changes in serum glucose and serum insulin concentrations between the intervention and placebo phases.

The Secondary outcomes include within-subject changes in:

* Lipid profile parameters: total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides, and the total cholesterol/HDL-c ratio.
* Anthropometric measurements: body weight, waist circumference, arm circumference, and body mass index (BMI).
* Blood pressure: systolic and diastolic, measured after rest.

Other Pre-specified Outcomes Glycemic control: Hemoglobin A1c (HbA1c).

* Liver and kidney function markers: including serum aspartate aminotransferase (AST), creatinine, and urea.
* Coagulation marker: Prothrombin time (PT).
* Complete blood count (CBC): including hemoglobin, white blood cell count, red blood cell count, and platelet count.
* Monitor systemic inflammatory status: Erythrocyte sedimentation rate (ESR)
* Adherence to the intervention (measured by portion tracking and consumption logs).
* Gastrointestinal symptom frequency (assessed via participant questionnaires).
* Product acceptability and palatability (evaluated using Likert-scale surveys).
* Participant-reported adverse events (monitored continuously throughout the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participant
* Men and women aged 20-59 years
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Documented food allergies, especially to legumes or beans
* Diagnosed liver, kidney, autoimmune diseases or severe illnesses such as cancer.
* Diagnosed gastrointestinal diseases including inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), celiac disease, or any condition causing chronic gastrointestinal symptoms such as malabsorption, persistent diarrhea, or gastrointestinal bleeding

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Glucose | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Venous blood samples will be collected at the beginning and end of each 4-week intervention phase to measure fasting serum glucose levels. The primary outcome is the within-subject difference in glucose concentration between the placebo and intervention periods. Values will be expressed in mg/dL.
Change in Serum Insulin | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Venous blood samples will be collected at the beginning and end of each 4-week intervention phase to measure fasting serum insulin levels. The primary outcome is the within-subject difference in insulin concentration between the placebo and intervention periods. Values will be expressed in µIU/mL.

SECONDARY OUTCOMES:
Change in Total Cholesterol | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Fasting serum total cholesterol will be measured at the beginning and end of each 4-week intervention phase. The outcome is the within-subject difference between the placebo and intervention periods. Values will be expressed in mg/dL.
Change in Triglycerides | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Fasting serum Triglycerides will be measured at the beginning and end of each 4-week intervention phase. The outcome is the within-subject difference between the placebo and intervention periods. Values will be expressed in mg/dL.
Change in HDL Cholesterol (HDL-c) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Fasting serum HDL-c will be measured at the beginning and end of each 4-week intervention phase. The outcome is the within-subject difference between the placebo and intervention periods. Values will be expressed in mg/dL.
Change in LDL Cholesterol (LDL-c) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Fasting serum LDL-c will be measured at the beginning and end of each 4-week intervention phase. The outcome is the within-subject difference between the placebo and intervention periods. Values will be expressed in mg/dL.
Change in Total Cholesterol to HDL-c Ratio | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  The ratio of total cholesterol to HDL-c will be calculated at baseline and after 4 weeks in each treatment period. The outcome is the within-subject difference between placebo and intervention. This value is unitless.
Change in Waist Circumference | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Waist circumference will be measured in centimeters using a non-elastic tape, to assess abdominal adiposity. The outcome is the within-subject difference between the placebo and intervention periods.
Change in Body Mass Index (BMI) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  BMI will be calculated using weight (kg) and height (m^2) at the beginning and end of each 4-week treatment period. Outcome will be expressed in kg/m^2 as the within-subject difference between placebo and intervention.
Change in Body Weight | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Body weight will be measured using a calibrated digital scale with participants wearing light clothing and no shoes. The outcome reflects the within-subject difference in weight between placebo and intervention phases. Values will be expressed in kilograms (kg).
Change in Blood Pressure (Systolic and Diastolic) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Blood pressure will be measured in mmHg after 5 minutes of rest, using a validated sphygmomanometer. Systolic and diastolic values will be recorded
Change in Arm Circumference | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Arm circumference will be measured in centimeters as a proxy for muscle or fat mass changes.

OTHER OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Fasting blood samples will be analyzed to determine the within-subject difference in HbA1c levels between placebo and intervention periods. Results will be expressed as a percentage (%).
Change in Serum Aspartate Aminotransferase (AST) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  AST will be measured to evaluate liver function and potential hepatic effects of the intervention. Units: U/L.
Change in Serum Creatinine | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Creatinine will be measured to assess renal function during the intervention. Units: mg/dL.
Change in Serum Urea (BUN) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Blood urea nitrogen will be assessed to monitor renal function. Units: mg/dL.
Change in Prothrombin Time (PT) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Prothrombin time will be measured to evaluate potential changes in coagulation. Results will be expressed in seconds and percentage (%).
Change in Hemoglobin Concentration | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Hemoglobin levels will be obtained from complete blood count (CBC) as an indicator of hematologic status. Units: g/dL.
Change in White Blood Cell Count (WBC) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  BC count will be analyzed as part of the complete blood count to monitor immune/inflammatory status. Units: numbers of cells x10^3/μL
Change in Red Blood Cell Count (RBC) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  RBC count will be analyzed as part of the complete blood count to monitor hematological status. Units: number of cells ×10^6/μL.
Gastrointestinal Symptom Frequency | Daily, during each 4-week treatment period.
  Participants will report gastrointestinal symptoms (e.g., bloating, gas, nausea, diarrhea) using a standardized weekly checklist. Frequency and severity will be described descriptively.
Adherence to Ice Cream Consumption Protocol | Throughout each 4-week phase (Week 0 and Week 4 of each treatment period)
  Adherence will be assessed by tracking the number of portions consumed compared to the number assigned. Results will be expressed as percentage of compliance.
Product Acceptability and Palatability | End of each 4-week treatment phase
  Acceptability of the ice cream will be evaluated through a 5-point Likert scale questionnaire covering taste, texture, and overall satisfaction. Results will be analyzed descriptively.
Participant-Reported Adverse Events | Continuous, during entire 8-week study period
  Any participant-reported adverse events will be recorded, including type, severity, and possible relationship with the intervention. Events will be categorized by frequency and seriousness.
Changes in Platelet Count | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Platelet count will be analyzed as part of the complete blood count to monitor hematological status and evaluate potential changes in platelet production or turnover. Units: number of cells ×10^3/μL
Change in Erythrocyte sedimentation rate (ESR) | Baseline and end of each 4-week phase (Week 0 and Week 4 of each treatment period)
  Erythrocyte sedimentation rate (ESR) will be analyzed to monitor systemic inflammatory status. Units: mm/hour

CONTACTS AND LOCATIONS:
Overall Officials: Ivan F Palomo González, PhD. Biomedical Science, Principal Investigator — University of Talca; Eduardo J Fuentes Quinteros, PhD. Science research, Principal Investigator — University of Talca
Locations (1):
- Universidad de Talca, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share individual participant data (IPD) has not yet been determined. The decision will depend on future publication plans, data management policies, and ethical considerations regarding participant privacy